CLINICAL TRIAL: NCT05003778
Title: The Effects of a Minimal Equipment Training Approach Compared to Concurrent Training to Improve Warfighter Health and Performance
Brief Title: Minimal Equipment Training Approach to Improve Warfighter Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Carolina (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Shawn M. Arent, Professor and Chair, University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00103649
Record Dates: First submitted 2021-07-21; First posted 2021-08-12 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Healthy; Military Operations
MeSH Terms: interventions — Blood Flow Restriction Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Traditional equipment resistance and endurance training (Active Comparator): Participants in this group undergo 6 weeks of concurrent resistance and endurance training using traditional equipment (i.e., power racks, barbells, dumbbells, etc.)
  Interventions: Other: Traditional equipment resistance training
- Minimal equipment resistance and endurance training (Experimental): Participants in this group undergo 6 weeks of concurrent resistance and endurance training using minimal equipment (i.e., sandbags, resistance bands, suspension trainers, weight vests, etc.)
  Interventions: Other: Minimal equipment resistance training
- Minimal equipment resistance and endurance training with blood flow restriction (Experimental): Participants in this group undergo 6 weeks of concurrent resistance and endurance training using minimal equipment (i.e., sandbags, resistance bands, suspension trainers, weight vests, etc.) while wearing upper- and lower-body blood-flow restriction cuffs
  Interventions: Other: Minimal equipment resistance training; Other: Blood flow restriction training

INTERVENTIONS:
Other: Traditional equipment resistance training — Participants will undergo 6 weeks of traditional equipment resistance training
  Arms: Traditional equipment resistance and endurance training
Other: Minimal equipment resistance training — Participants will undergo 6 weeks of minimal equipment resistance training
  Arms: Minimal equipment resistance and endurance training; Minimal equipment resistance and endurance training with blood flow restriction
Other: Blood flow restriction training — Participants will undergo 6 weeks of blood flow restriction training
  Arms: Minimal equipment resistance and endurance training with blood flow restriction

SUMMARY:
The purpose of this project is to compare a minimal equipment training program with and without blood flow restriction (BFR) training to periodized concurrent resistance and endurance training. The outcomes of interest are Army Combat Fitness Test (ACFT) performance along with laboratory measures of performance, which include body composition, power, strength, and maximal aerobic capacity (VO2max). Additionally, based on the role of mechanical tension in connective tissue adaptation and the importance for chronic musculoskeletal health, tendon architecture will be assessed as well. Lastly, specific blood-based biomarkers will be analyzed in conjunction with questionnaires to determine the systemic physiological and psychological responses to training. Participants will be randomized into one of three training groups and will follow their respective program for 6 weeks. The three groups are traditional concurrent resistance and endurance training, minimal equipment training, and minimal equipment training with blood flow restriction (BFR).

DETAILED DESCRIPTION:
The efficacy of minimal equipment training programs with an emphasis on resistance training has seldom been assessed and compared to traditional strength training. Common training strategies include traditional high-to-moderate load resistance training and low-to-moderate load field training using minimal equipment. The benefit of traditional CT is likely due to the higher loads relative to 1-repetition maximum (1RM) utilized and overall amount of mechanical stress incurred. It is difficult to mimic this loading with minimal equipment training, which is often performed at low loads relative to 1RM. However, one strategy to improve the effectiveness of minimal equipment training may be the addition of blood flow restriction (BFR) training. Due to the relatively low loads (20-70% 1RM) of minimal equipment training, BFR training not only provides athletes with a novel training modality to elicit hypertrophic and strength adaptation but also to augment recovery as a supplemental low-damage, high-volume training method. The research design will allow for the direct comparison of minimal equipment training with and without additional BFR training to periodized CT with regard to changes in outcomes, in particular, ACFT performance.

ELIGIBILITY:
Inclusion Criteria:

* Males and females between the ages of 18 and 35 (inclusive) and enrolled in an ROTC program.
* Subject has provided written and dated informed consent to participate in the study.
* Subject is in good health as determined by medical history and is cleared for exercise.
* Subject will be asked about dietary supplementation use within the past 6 months.

  * If subject began taking a supplement within the past month, subject will be asked to discontinue supplement use followed by a 2-week washout prior to participation.
  * In all other cases, we will request that subjects maintain supplement use.

Exclusion Criteria:

* Subjects with any musculoskeletal injuries that would prevent exercising.
* Subjects with any metabolic disorder including known electrolyte abnormalities, diabetes, thyroid disease, adrenal disease or hypogonadism.
* Subjects with any inborn error of metabolism.
* Subjects with a history of hepatorenal, musculoskeletal, autoimmune, or neurologic disease.
* Subjects with a personal history of heart disease, high blood pressure (systolic >140 mm Hg & diastolic >90 mm Hg), psychiatric disorders, cancer, benign prostate hypertrophy, gastric ulcer, reflux disease, or any other medical condition deemed ineligible to participate in physical training by the ROTC athletic trainers or ROTC medical staff.
* Subjects currently taking thyroid, hyperlipidemic, hypoglycemic, anti-hypertensive, or anti-coagulant medications.
* Subjects who are pregnant or lactating.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2020-11-20 (Actual); Primary Completion 2022-03-04 (Actual); Study Completion 2022-06-29 (Actual)

PRIMARY OUTCOMES:
Change in Army Combat Fitness Test | Baseline and Week 6
  6-event task to assess various aspects of human performance (muscular power, muscular strength, muscular endurance, anaerobic capacity, and aerobic capacity). Tests include 3-repetition maximum trap-bar deadlift, standing power throw with 10-lb ball, 2-min hand-release push-ups, sprint-drag-carry, 2-min leg tucks, and 2-mile run.

SECONDARY OUTCOMES:
Change in muscular power | Baseline and Week 6
  Assessed via countermovement vertical jump height.
Change in muscular strength | Baseline and Week 6
  Assessed via 3-repetition maximum bench press.
Change in aerobic capacity | Baseline and Week 6
  Assessed via treadmill-based maximal graded exercise test with indirect calorimetry.
Change in body mass | Baseline and Week 6
  Body mass via calibrated scale.
Change in body composition | Baseline and Week 6
  Body fat percentage, fat-free mass, and fat mass via air-displacement plethysmography.
Change in muscle and tendon thickness | Baseline and Week 6
  Biceps brachii and quadriceps muscle thickness via B-mode ultrasound and distal biceps tendon and quadriceps tendon via B-mode ultrasound.
Change in blood-based biomarkers | Baseline and Week 6
  Basal hormonal and biochemical assessments. Cortisol, interleukin (IL)-6, IL-10, IL-1β, growth hormone (GH), and insulin-like growth factor-1 (IGF-1).
Change in blood lactate responses | Baseline, Week 3, and Week 6
  Biochemical responses to exercise. Blood lactate sampled pre-, mid-, and post-exercise during training sessions in weeks 1, 3, and 6.
Change in training distress | Baseline and every subsequent week through Week 6
  Overall training distress and subscales including depressed moods, vigor, physical signs and symptoms, sleep disturbances, perceived stress, and general fatigue. The Multicomponent Training Distress Scale will be administered weekly.

CONTACTS AND LOCATIONS:
Locations (1):
- University of South Carolina Sport Science Lab, Columbia, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cintineo HP, Chandler AJ, Mastrofini GF, Lints BS, McFadden BA, Arent SM. Effects of Minimal-Equipment Resistance Training and Blood Flow Restriction on Military-Relevant Performance Outcomes. J Strength Cond Res. 2024 Jan 1;38(1):55-65. doi: 10.1519/JSC.0000000000004596. PMID 38085621